CLINICAL TRIAL: NCT06543888
Title: Effects of Passive Lower-limb Exoskeleton-assisted Training on Motor and Daily Function Improvements in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 202302129B0
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Multidomain Intervention
Keywords: aging; motor function,; gait,; exoskeleton

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- passive exoskeleton- assisted gait training programs (Experimental): Behavioral: passive exoskeleton- assisted gait training programs Participants will receive 12 sessions of passive exoskeleton-assisted gait training programs (30 min/session, 3 sessions/week for 4 consecutive weeks).
  Interventions: Behavioral: passive exoskeleton- assisted gait training programs
- conventional gait training programs (Active Comparator): Participants will receive 12 sessions of conventional gait training programs (30 min/session, 3 sessions/week for 4 consecutive weeks).
  Interventions: Behavioral: Conventional gait training

INTERVENTIONS:
Behavioral: passive exoskeleton- assisted gait training programs — Participants will wear an exoskeleton during the training. Each 30-minute Passive exoskeleton-assisted gait training session include range of motion exercise, movement facilitation, strengthening exercise, coordination exercise, and task-oriented training for activities of daily living
  Arms: passive exoskeleton- assisted gait training programs
Behavioral: Conventional gait training — Each 30-minute conventional gait training session include range of motion exercise, movement facilitation, strengthening exercise, coordination exercise, and task-oriented training for activities of daily living.
  Arms: conventional gait training programs

SUMMARY:
According to National Development Council estimation, Taiwan is about to enter a super-aged society in 2025, and health promotion for the elderly are critical issues nowadays. The age-related decline in motor function will further affect participation in activities of daily living. In addition to conventional rehabilitation training, robot-assisted training has gained acceptance in clinical rehabilitation. However, robot-assisted trainings were mostly used for motor recovery in patients with neurological disorders, and has not yet been applied to motor function training in community dwelling older adults. This study will examine the effect of passive exoskeleton-assisted gait training on motor function, daily function and self- efficacy in community dwelling older adults, so as to achieve health promotion and develop a new training approach. The purpose of this study will be to determine the comparative effects of passive exoskeleton-assisted gait training and conventional gait training on motor and daily function improvements in older adults.

ELIGIBILITY:
Inclusion Criteria:

1. age ≧ 60
2. normal functional range of motion (within functional limits) in trunk, and leg joints
3. ability to walk continuously for 10 minutes with or without an assistive device
4. Mini Mental State Exam (MMSE) score > 24, indicating no serious cognitive impairment

Exclusion Criteria:

1. histories of neurological diseases such as dementia, Parkinson's disease, and peripheral polyneuropathy
2. recent lower leg injury (6 months) or surgery (1 year) based on self-report
3. taking any over-the-counter drugs, prescription medications, or any substance that may affect gait
4. difficulties in following and understanding instructions
5. enroll in other rehabilitation or drug studies simultaneously -

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-03-17 (Estimated); Study Completion 2027-03-17 (Estimated)

PRIMARY OUTCOMES:
Change scores of Five Times Sit to Stand Test (FTSST) | Baseline, post test after completing 12 intervention sessions (around 4 weeks after baseline), follow up test (1 month after completing intervention sessions)]
  The FTSST measures the time taken to stand five times from a sitting position as fast as possible, which is used to assess functional lower limb strength, balance control, and mobility in both healthy adults and those with pathologies. The FTSST has been proven to be safe and to have excellent reliability.
Change scores of Timed Up and Go Test (TUG) | Baseline, post test after completing 12 intervention sessions (around 4 weeks after baseline), follow up test (1 month after completing intervention sessions)]
  The TUG test assesses dynamic balance ability and mobility. The participants will be required to stand up from a chair, walk 3 m, turn around, walk back to the chair, and sit down. Three trials will be taken at each assessment, and the average of three trials will be documented. The time to complete the TUG test has been shown to be a good indicator to detect potential fallers in frail elderly individuals. The TUG is a reliable, valid, and easy-to-administer clinical tool.
Change scores of 10-meter walk test (10MWT) | Baseline, post test after completing 12 intervention sessions (around 4 weeks after baseline), follow up test (1 month after completing intervention sessions)]
  The 10MWT assesses walking speed in self-selected pace and fast walking pace, which can be employed to determine functional mobility. Two trials are administered at the participant's comfortable walking speed, followed by 2 trials at his/her fast walking speed. The 2 trials, for each speed, are averaged and the 2 gait speeds are documented in meters/second. The 10-meter walk test has demonstrated excellent
  reliability for comfortable and fastest gait speeds in healthy adults and other pathological populations.
Change scores of Nottingham Extended Activities of Daily Living Scale (NEADL) | Baseline, post test after completing 12 intervention sessions (around 4 weeks after baseline), follow up test (1 month after completing intervention sessions)]
  The NEADL is a measure of independence in 4 areas of daily life, including mobility, kitchen, domestic, and leisure activities. It includes 22 items, and each item is measured on a 4-point scale. The total score ranges from 0 to 66 and a higher score indicates better daily functional ability. The psychometric properties of the NEADL have been well established.
Change scores of Daily Living Self-Efficacy Scale (DLSES) | Baseline, post test after completing 12 intervention sessions (around 4 weeks after baseline), follow up test (1 month after completing intervention sessions)]
  The DLSES measures self-efficacy of daily functioning, including psychosocial functioning and activities of daily living. The scale consists of 12 items, and each item is measured on a 100-point scale with 10-unit intervals (0 = cannot do at all, 100 = highly certain can do). A higher score indicates higher level of self-efficacy. The DLSES is a psychometrically sound measure of self-efficacy in stroke survivors.
Change scores of Functional Abilities Confidence Scale (FACS) | Baseline, post test after completing 12 intervention sessions (around 4 weeks after baseline), follow up test (1 month after completing intervention sessions)]
  The FACS measures the degree of self-efficacy and confidence when the participants perform various movements and postures. It consists of 15 questions scoring from 0% (not confidence at all) to 100% (fully confidence). A higher score indicates higher confidence of performing the movements. The psychometric properties are good.
Change scores of Mini-Mental State Examination (MMSE) | Baseline, post test after completing 12 intervention sessions (around 4 weeks after baseline), follow up test (1 month after completing intervention sessions)]
  The MMSE a 30-point questionnaire that is the most commonly used brief screening tool for detecting cognitive impairment. Higher values represent a better cognitive functioning. The MMSE has good psychometric properties for identifying cognitive impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memotial Hospital, Taoyuan District, Guishan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided